CLINICAL TRIAL: NCT06116396
Title: Use of Urinary Tumor Cells and Circulating Tumor Cells (CTCs) in the Prognosis and Therapy of Patients With Bladder (BCa) and Upper Urinary Tract (UTUC) Cancer"
Brief Title: Liquid Biospy for Urinary Cancers
Acronym: CIRCE
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Alfano, PhD, IRCCS San Raffaele
Other Study IDs: CIRCE
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Urothelial neoplasia
  Interventions: Genetic: Genetic analysis on isolated cells
- 2: Age-matched individuals free of neoplasia
  Interventions: Genetic: Genetic analysis on isolated cells

INTERVENTIONS:
Genetic: Genetic analysis on isolated cells — Isolation of cells from blood and urine

SUMMARY:
The project aims to characterize the prognostic role of CTCs in Bladder cancer patients, with the specific aims to better stratify patients with non-muscle invasive bladder cancer at the first transurethral resection of tumor and to identify urothelial biomarker expressed by CTCs.

DETAILED DESCRIPTION:
Bladder cancer (BCa) is the 9th most common cancer worldwide, with an estimated prevalence of around 2.7 million cases and an incidence around 350.000 new cases/year. The proper management of BCa remains an unmet clinical need, because one of the main problems in BCa treatment is the inability to efficaciously prevent high-grade non-muscle invasive bladder cancer (NMIBC) relapse and progression, which occur in 80% and 45% of patients respectively. Indeed, as a consequence of the lack of efficient established prognostic, diagnostic and predictive biomarker of high-risk NMIBC, Bca patients undergo multiple treatments and cystoscopic assessments along their life, with consequent poor quality of life and high healthcare costs.

Circulating Tumor Cells (CTCs) in blood represent an invaluable source of tumor material that can be easily collected yhrough a simple blood draw and may represent the clonal component of the primary tumor that left the primary site.

For this reason, the aim of this study is to characterize the prognostic role of CTCs in Bladder cancer patients, with the specific aims to better stratify patients with non-muscle invasive bladder cancer at the first transurethral resection of tumor and to identify urothelial biomarker expressed by CTCs.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of urothelial neoplasia, naive for therapy

Exclusion Criteria:

Absence of previous neolpastic disease or genetic diseases

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults men and women.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of the liquid biopsy | 2020-2023
  Gene signature in CTC and UTC predicting tumor relapse

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Alfano, PhD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- Urology Department, Milan, Italy